CLINICAL TRIAL: NCT01601652
Title: Open Label, Compassionate Use Protocol of an Intravenous Fish Oil Emulsion in Infants With Cholestasis
Brief Title: Compassionate Use of an Intravenous Fish Oil Emulsion in Infants With Cholestasis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Arthur J De Lorimier (Other)
Responsible Party: Sponsor-Investigator, Arthur J De Lorimier, Associate Professor of Pediatrics, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 225576; UCD#225576-3 (Other: UC Davis)
Record Dates: First submitted 2012-05-09; First posted 2012-05-18 (Estimated); Results first posted 2021-01-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Parenteral Nutrition Associated Cholestasis
Keywords: cholestasis; PNAC; Parenteral Nutrition Associated Cholestasis; PNALD; Parenteral Nutrition Associated Liver Disease
MeSH Terms: conditions — Cholestasis | interventions — fish oil triglycerides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Omeagven (Experimental)
  Interventions: Drug: Omegaven

INTERVENTIONS:
Drug: Omegaven — 1 g/kg/d iv infusion over 24h

SUMMARY:
The study will evaluate the safety and efficacy of an intravenous fish oil emulsion (omegaven) in infants with parenteral nutrition associated cholestasis.

ELIGIBILITY:
Inclusion Criteria:

Cholestasis defined as either

* serum bilirubin > 2mg/dL (two measurements at least 8d apart) that has not responded to 4 weeks of intralipid being reduced to 1 g/kg/d and trace minerals being limited to twice weekly, OR
* serum bilirubin > 6 mg/dL (single measurement) and rising, in the absence of proven or suspected sepsis

Exclusion Criteria:

* Age > 1y at time that omegaven is started
* Not expected to survive at least 30 days
* Fish allergy in a first degree relative
* Hemodynamic instability
* Coagulopathy
* Not likely to require PN for > 30d
* Not expected to survive > 30d

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2011-11; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian J Griffin, MD, Principal Investigator — UC Davis
Locations (1):
- University of California Davis Medical Center, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Started Omegaven: N=12
  1 Died of complications not related to omegavin 5 Weaned off PN before DC (2F, 3M) 6 Discharged Home on PN (of these 3 remain on PN[all male]; 3 weaned off after DC [2M, 1F])
Period: Overall Study
Arm/Group | Omeagven
Started (12 started omegaven 1 Died of complications unrelated to omegaven 6 DC home on PN (3M still on PN; 2M & 1F weaned from PN) 5 Weaned from PN prior to DC (2F, 3M)) | 12
Completed (Last patient admitted to study on 2/18/2017 and data collection ended a month later.) | 11
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: 12 started omegaven
  1 Died M 5 weaned off PN in NICU (2F, 3M) 6 DC home on PN (3M continue on PN; 2M &1F weaned off )
Arm/Group | Omeagven
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: month] | 10 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Normalization of Conjugated Bilirubin (Conjugated Bilirubin < 2 mg/dL)
Time Frame: approximately for 4 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Omeagven
Number analyzed (Participants) | 11
mg/dl | 2 (0.2)

2. Secondary Outcome: Liver Transaminases
Time Frame: approximately for 4 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Omeagven
Number analyzed (Participants) | 11
mg/dl | 98 (10)

ADVERSE EVENTS:
Time Frame: 36 mo
Arm/Group | Omeagven
All-Cause Mortality (participants affected / at risk) | 1/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omeagven (N=12)
hypertriglyceridemia (Gastrointestinal disorders) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-01-12): https://cdn.clinicaltrials.gov/large-docs/52/NCT01601652/Prot_SAP_000.pdf
  • Informed Consent Form (2018-02-12): https://cdn.clinicaltrials.gov/large-docs/52/NCT01601652/ICF_001.pdf